CLINICAL TRIAL: NCT05865639
Title: Effects of Time Restricted Fasting and Exercise on Cardiovascular Risks Among Sedentary Adults
Brief Title: Time Restricted Fasting and Aerobic Exercise Interventions Among Sedentary Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Sport University (Other)
Collaborators: Guangdong Provincial Key Laboratory of Physical Activity and Health Promotion (Unknown); Guangdong Provincial Scientific Research Center (Unknown)
Responsible Party: Principal Investigator, Jingwen Liao, Associate Professor, Guangzhou Sport University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20230411
Record Dates: First submitted 2023-04-13; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Sedentary; Aging
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic Exercise (Experimental): Aerobic exercise for eight weeks. Three weekly, supervised training sessions.
  Interventions: Behavioral: Aerobic Exercise
- Time Restricted Fasting (Experimental): Time restricted fasting for eight weeks. Maximal daily eating window of 8 hours.
  Interventions: Behavioral: Time Restricted Fasting
- Aerobic exercise & Time Restricted Fasting (Experimental)
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Time Restricted Fasting
- Control (No Intervention): Will be given information about the recommended level of physical activity for health benefits and a healthy diet.

INTERVENTIONS:
Behavioral: Aerobic Exercise — Three weekly, supervised exercise sessions with aerobic exercise. Each session will last for 60-65 minutes, each period will be consist of 5 min warm up, 45 min formal training and 5-10 min relaxation training. Intervention period will be eight weeks.
  Arms: Aerobic Exercise; Aerobic exercise & Time Restricted Fasting
Behavioral: Time Restricted Fasting — Restricted daily window of caloric intake to maximum 8 hours. Intervention period will be eight weeks.
  Arms: Aerobic exercise & Time Restricted Fasting; Time Restricted Fasting

SUMMARY:
This project will determine the independent and combined effects of aerobic exercise and time restricted fasting on cardiovascular risks among sedentary middle-aged and elderly adults. The online intervention period will be eight weeks. Before and after the intervention, arterial stiffness, cardiac autonomic nervous, body composition, glucolipid metabolism, sleep and eating habits, inflammatory reaction, sedentary behavior and physical activity level will be measured and compared between groups who are doing either aerobic exercise, time restricted fasting, both aerobic exercise and time restricted fasting, or who are in a control group. Adverse reaction, sleep and eating quality, life quality and adherence to the interventions and hunger/satiety will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45-69 years old Sedentary time ≥8 hours per day
* Irregular exercise habits
* No drugs affecting the outcome index were taken
* No history of serious diseases
* Sign the subject informed consent and agree to participate in this experiment.

Exclusion Criteria:

* The range of body weight change in the last three months is more than 3kg
* People taking weight-loss drugs
* Participate in other experimenters 5 months before the experiment
* Unable to adjust and follow the intervention schedule.

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change of cardiovascular risk estimated by heart rate variability | From baseline to after 8 weeks intervention
Change of cardiovascular risk estimated by ankle-brachial index | From baseline to after 8 weeks intervention
Change of cardiovascular risk estimated by pulse wave velocity | From baseline to after 8 weeks intervention
Change of cardiovascular risk estimated by flow-mediated transition | From baseline to after 8 weeks intervention
Change of cardiovascular risk estimated by cytokines level | From baseline to after 8 weeks intervention
  Fasting matrix metalloproteinases, norepinephrine, and neuropeptide Y cytokines level in blood

SECONDARY OUTCOMES:
Weight | From baseline to after 8 weeks intervention
  In kg
body fat | From baseline to after 8 weeks intervention
  In kg
Lean body mass | From baseline to after 8 weeks intervention
  In kg
Body mass Index | From baseline to after 8 weeks intervention
  In kg/m^2
Body fat percentage | From baseline to after 8 weeks intervention
  In percent of total body mass
Diet habits | From baseline to after 8 weeks intervention
  Self-reported: diet habits were assessed using the Adult Eating Behavior Questionnaire (AEBQ).
  With higher scores indicating worse eating habits (represented by emotional over-eating and emotional under-eating) or better dietary (represented by food responsiveness, enjoyment of food, satiety responsiveness, food fussiness and slowness in eating).
Sleep quality | From baseline to after 8 weeks intervention
  Self-reported: sleep quality was indicated by the Pittsburgh Sleep Quality Index (PSQI) Questionnaire. The maximum score of the sleep quality index is 21 points,scores higher than 5 indicate poor sleep quality, with higher scores indicating poorer sleep quality.
Life quality | From baseline to after 8 weeks intervention
  Self-reported: life quality was indicated by The World Health Organization Quality of Life (WHOQOL)-BREF Questionnaire. With higher scores indicating better life quality.
Physical activity | From baseline to after 8 weeks intervention
  Physical activity were measured by using accelerometer (ActiGraph GT3X+ model, USA).Measured by using accelerometer (ActiGraph GT3X+ model, USA). Accelerometer was used for 7 consecutive days, being affixed to the nondominant wrist.
Sedentary activity | From baseline to after 8 weeks intervention
  Sedentary activity were measured by using accelerometer (ActiGraph GT3X+ model, USA).Measured by using accelerometer (ActiGraph GT3X+ model, USA). Accelerometer was used for 7 consecutive days, being affixed to the nondominant wrist.
Inflammation level | From baseline to after 8 weeks intervention
  Inflammation level were measured by Enzyme-linked immuno sorbent.
Cholesterol in blood | From baseline to after 8 weeks intervention
  Total fasting cholesterol in blood
High density lipoprotein in blood | From baseline to after 8 weeks intervention
  Fasting high density lipoprotein in blood
Low density lipoprotein in blood | From baseline to after 8 weeks intervention
  Fasting low density lipoprotein in blood
Triglycerides in blood | From baseline to after 8 weeks intervention
  Fasting triglycerides in blood
Diet in take | From baseline to after 8 weeks intervention
  Self-reported: Mint Health application.
Adherence to intervention | From baseline to after 8 weeks intervention
  Self-reported: WeChat application, number of completed exercise sessions out of those prescribed, in percentage.
Adverse reaction | From baseline to after 8 weeks intervention
  Self-reported: mini program.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Sport University, Guangdong, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No